CLINICAL TRIAL: NCT04628520
Title: Effect of Soft Tissue Augmentation Procedures on Peri-implant Health
Brief Title: Surgical Protocol for Prevention of Mucositis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Clementini, Principal Investigator, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mucositis surgical
Record Dates: First submitted 2020-10-31; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Mucositis
Keywords: CTG; Mucositis; Surgical Treatment; Keratinised tissue; Free gingival graft; Collagen matrix
MeSH Terms: conditions — Mucositis | interventions — Maintenance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Maintenance (Sham Comparator): Oral hygiene instruction and periodontal maintenance
  Interventions: Procedure: Maintenance
- Free gingival graft (Active Comparator): After administration of local anesthesia, an intrasulcular incision will be made at the muco-gingival line and a partial thickness flap will be raised and sutured at the base of the newly created vestibule with resorbable mattress sutures. After the completion of the apically positioned flap, patients will receive a free gingival graft (FGG) harvested from the palate, that will be fixed with interrupted resorbable sutures to the recipient periosteal bed, free of any muscle attachment.
  Interventions: Procedure: Free gingival graft; Procedure: Maintenance
- Collagen matrix (Active Comparator): After administration of local anesthesia, an intrasulcular incision will be made at the muco-gingival line and a partial thickness flap will be raised and sutured at the base of the newly created vestibule with resorbable mattress sutures. After the completion of the apically positioned flap, patients will receive either a collagen matrix (CM), that will be fixed with interrupted resorbable sutures to the recipient periosteal bed, free of any muscle attachment.
  Interventions: Procedure: Collagen matrix; Procedure: Maintenance

INTERVENTIONS:
Procedure: Free gingival graft — After administration of local anesthesia, an intrasulcular incision will be made at the muco-gingival line and a partial thickness flap will be raised and sutured at the base of the newly created vestibule with resorbable mattress sutures. After the completion of the apically positioned flap, patients will receive a free gingival graft (FGG) harvested from the palate, that will be fixed with interrupted resorbable sutures to the recipient periosteal bed, free of any muscle attachment.
  Arms: Free gingival graft
Procedure: Collagen matrix — After administration of local anesthesia, an intrasulcular incision will be made at the muco-gingival line and a partial thickness flap will be raised and sutured at the base of the newly created vestibule with resorbable mattress sutures. After the completion of the apically positioned flap, patients will receive either a collagen matrix (CM), that will be fixed with interrupted resorbable sutures to the recipient periosteal bed, free of any muscle attachment.
  Arms: Collagen matrix
Procedure: Maintenance — Oral Hygiene Instruction, periodontal debridment and Supportive Periodontal Therapy

SUMMARY:
The main goal of implant therapy is to obtain long-term peri-implant health. Among local risk factors in the etiology of peri-implant diseases the absence of keratinized tissue (KT) around the implant has been reported. In fact, a certain amount of KT width, providing better sensory isolation and, hence, less pain discomfort during brushing, may be useful to facilitate plaque control. A good plaque control should maintain periimplant health during time.

A very recent systematic review assessed the effect of soft tissue grafting procedures on peri-implant health, revealing that soft tissue grafting using autogenous tissue for gain of KT results in a significant decrease of PI, BOP and GI values and significantly lower PI and GI values and higher marginal bone levels at the study endpoint compared to maintenance groups.

DETAILED DESCRIPTION:
Based in the available data in literature, it has been demonstrated that the level of brushing discomfort was significantly higher in sites with <2 mm of KT width, which exhibited more plaque and more bleeding on probing than sites with ≥2 mm of KT width. Therefore, various procedures and materials were proposed in the past to augment the soft tissues around dental implant. Soft-tissue grafting seems beneficial, especially in posterior mandible, when patients complains of soreness during oral hygiene procedures and plaque control is less than ideal and it may be facilitated by a better topography. The surgical procedures most frequently used to increase the width of keratinized tissue around an implant-supported restoration include an apically positioned split-flap/vestibuloplasty (APF) with or without the application of autogenous tissue (i.e., free gingival graft) or a xenogeneic collagen matrix.

However, it remains unclear whether or not surgical procedures for gain of KT may establish peri-implant health limiting the incidence of peri-implant disease and may positively affect self-performed oral hygiene measures reducing peri-implant soft tissue inflammation when compared with non-augmented, inadequately dimensioned implant sites. Neither do clinical suggestions exist for a specific soft tissue transplant to obtain more favorable outcomes.

The aim of the present randomized controlled clinical trial is to assess the effect of soft tissue augmentation procedures at diseased (mucositis) implant sites in terms of:

* occurrence of peri-implant health (absence of BoP/suppuration, PPD>6mm, longitudinal radiographic bone loss) at 3, 6 and 12 months
* reduction of BoP (%) at 3, 6 and 12 months
* marginal bone loss (MBL) at 12 months
* improvement of self-performed oral hygiene measures (PI, VAS) at 3, 6 and 12 months and post-operative morbidity (VAS) at 7 days.
* change in tissue morphology: increase of KT width (2D in mm.) and tissue volume (volumetric 3D) at 3, 6 and 12 months and aesthetic (blinder examiner) at 6, 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Systemic healthy patients
* appropriate oral hygiene standards (full mouth plaque scores <20%)
* periodontal health (BoP < 10%) or gingivitis (BoP > 10%) in a healthy or reduced periodontium
* clinical signs of mucositis (presence of BoP) at the affected implant-supported fixed prosthesis
* < 2mm of KT at the mid-buccal aspect of implant-supported fixed prosthesis
* < 10 cigarette/die

Exclusion Criteria:

* any systemic disease that would negatively influence wound healing or known allergy to collagen
* more than 10 cigarettes/day
* sites with implant-supported rehabilitations presenting poor marginal adaptation (confirmed by an explorative probe and radiographic examination)
* implant-supported rehabilitations with inadequate access to hygiene

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
peri-implant health occurrence | 6 and 12 months after treatment
  percentages of clinical cases with the following characteristics for each treated implant: absence of Bleeding on Probing (BoP), Probing Pocket Depth (PPD) <6mm, absence of marginal bone loss (MBL)

SECONDARY OUTCOMES:
Bleeding on probing (BoP) changes | 3, 6 and 12 months after treatment
  changes of bleeding on probing, evaluated as present if bleeding will be evident within 15 s after gentle probing, or absent, if no bleeding will be noticed within 15 s after probing
Plaque index (PI) changes | 3, 6 and 12 months after treatment
  changes in plaque index, evaluated as present if identifiable plaque will be evident, with the use of a periodontal probe along the gingival margin, or absent, if no plaque will be noticed
Probing pocket depth (PPD) changes | 3, 6 and 12 months after treatment
  changes in probing pocket depth, assessed from the peri-implant mucosa margin to the the bottom of the peri-implant sulcus, measured in millimeters
mucosal recession (REC) changes | 3, 6 and 12 months after treatment
  changes in mucosal recession, assessed from the implant shoulder to the peri-implant mucosa margin, measured in millimeters
Keratinized tissue changes ( KT) | 3, 6 and 12 months after treatment
  width of KT, assessed from the gingival margin to the mucogingival junction at the mid-buccal aspect of the implant measured through "rolling technique" in millimeters
marginal bone loss (MBL) | 6 and 12 months after treatment
  marginal bone loss at mesial and distal aspect, measured on periapical X-ray
discomfort during oral hygiene procedure | baseline, 3, 6 and 12 months after treatment
  the level of brushing discomfort experienced by patients during oral hygiene will be evaluated, using a 0 to 100 mm visual analog scale (VAS). Patients will be invited to mark a point in the line that will represent the level of discomfort they felt during the brushing procedure, varying from 0 (no discomfort) to 100 (extreme discomfort).
post-surgical morbidity | 7 days after treatment
  the level of post-operative morbidity will be evaluated through a 0 to 100 mm visual analog scale (VAS) and the amount of anti-inflammatory medication used by the patient. The investigator will record the presence of complications, additional treatments, and medication in connection to the surgical treatment, using a specific form and a questionnaire handed to the patients.
volumetric changes | 3, 6 and 12 months after treatment
  digital impressions will be obtained using a 3D scanner in order to create stereolithography (STL) files. STL files of each patient will be superimposed and matched using a digital volume comparison software program. Superimposed STL files will be used to assess linear and volumetric soft tissue dimensional changes (linear and volumetric soft tissue contour changes).
aesthetic | 6 and 12 months after treatment
  aesthetic will be evaluated by a blinder examiner with the pink esthetic score (PES) as described by Fürhauser et al. 2005

CONTACTS AND LOCATIONS:
Overall Officials: Massimo De Sanctis, Study Chair — Università Vita-Salute San Raffaele
Locations (1):
- Università Vita-Salute San Raffaele, Milan, Italy